CLINICAL TRIAL: NCT00138294
Title: Phase 4, School-based, Open-labeled Research Trial for Control of Epidemic Influenza Through a School-based Influenza Vaccination Program in Central Texas.
Brief Title: Control of Epidemic Influenza Through a School-based Influenza Vaccination Program
Acronym: CEI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Scott and White Hospital & Clinic (Other); Novartis (Industry); Sanofi Pasteur, a Sanofi Company (Industry); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Pedro Piedra, Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BCM H-21853; Flu-035-09 (Other: MedImmune Inc); BCM H-21853 (Other: Baylor College of Medicine); SW070912 (Other: Scott and White); R01AI041050 (NIH)
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Influenza
Keywords: influenza vaccine; live attenuated influenza vaccine (LAIV or FluMist); inactivated influenza vaccine (IIV); School-based influenza vaccination program; children; herd protection
MeSH Terms: conditions — Influenza, Human | interventions — FluMist; Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Cities (Experimental): Children 4 years of age and older in the intervention cites (Temple, Belton, Academy, Troy, Salado, Rogers, and Holland) with be offered live attenuated or inactivated influenza vaccines through a school-based research vaccination program.
  Interventions: Biological: live attenuated and inactivated influenza vaccines
- Comparison Cities (Active Comparator): Children living in the comparison cities (Waco, Bryan and College Station) which are within 90 miles of the intervention cites will received their influenza vaccines (live attenuated or inactivated influenza vaccines) by the local healthcare providers.
  Interventions: Biological: live attenuated and inactivated influenza vaccines

INTERVENTIONS:
Biological: live attenuated and inactivated influenza vaccines — Live Attenuated Influenza Vaccine (LAIV) and Inactivated Influenza Vaccine (IIV) were administered to eligible children through a research program to improve vaccination coverage in school-aged children. Children 4 years of age and older in the intervention cites (Temple, Belton, Academy, Troy, Salado, Rogers, and Holland) will be offered LAIV or IIV through a school-based research vaccination program. Children living in the comparison cities (Waco, Bryan and College Station) which are within 90 miles of the intervention cites received LAIV or IIV from the local healthcare providers
  Other Names: FluMist; Fluzone

SUMMARY:
The main purpose of this study is to learn if influenza vaccines (live attenuated and inactivated influenza vaccines), when given to school-aged children 4 to 18 years of age, can stop or lessen the influenza (flu) outbreak in the community. Another purpose is to show that vaccination of these children will significantly reduce breathing problems (in the vaccinated children and unvaccinated people they come in contact with in the community) that require a visit to the doctor for treatment. Another purpose is to continue to collect safety and flu protection information on live attenuated influenza vaccine (LAIV or FluMist) given to children. The study investigators believe that vaccination of healthy school-aged children is an effective plan for preventing many people in the community from catching the flu. Children will take part in the study for 5 to 10 months.

DETAILED DESCRIPTION:
This study was conducted in three phases. The first phase spanned from 1998-2003 (PubMed ID:14706961; PubMed ID: 12915495) and the second phase spanned from 2003-2007 (PubMedID: 18401289; PubMed ID: 17698577). The final phase of the study spanned 2007-2011 and is the scope of this submission.

The goal of the final phase is to control epidemic influenza through active immunization of healthy school-aged children with the cold-adapted, trivalent, live, attenuated influenza vaccine (LAIV) and at-risk children with the inactivated influenza vaccine (IIV) through a school-based vaccination program.

The hypothesis is that universal vaccination of healthy school-aged children is an alternative and effective strategy for the control of epidemic influenza, and will serve as a model for the control of pandemic influenza and biodefense. The specific aims of the study are: to control the spread of influenza to susceptible adults 35 years of age or older by vaccination of school-aged children 4-18 years of age; to control the spread of influenza to susceptible children and young adults less than 35 years of age by vaccination of school-aged children 4-18 years of age; to develop a school-based vaccination program for rapid and timely delivery of LAIV and IIV to children 4-18 years of age; to demonstrate in school-aged children the direct and total effectiveness of influenza vaccines to reduce the rates of medically attended acute respiratory illness (MAARI) in LAIV and IIV recipients during influenza epidemics; and to capture safety information on LAIV post-licensure.

This is an open-label, up to four year community-based study. In each of the first three study years, school-aged children (4 through 18 years of age) who receive medical care at the Scott & White Clinics (SWCs), Temple-Belton area, Texas, will be asked to participate in this study. Study participants will receive LAIV or IIV according to their health status. Other children from Temple-Belton area who do not receive medical care at the SWC will be invited to participate in the study and may receive LAIV or IIV. A comparable population enrolled in the SWCs in Waco/McLennan County area and Bryan/College Station will serve as comparison groups.

In the fourth and final year of the study, LAIV will not be provided through the study. However, influenza surveillance will continue and MAARI data will be collected to assess continued protective benefit of influenza vaccines. The final year will also be devoted to completion of data analysis and preparation of manuscripts.

Children 4 years through 8 years who have not previously been vaccinated with an influenza vaccine will be offered a second dose 4 to 6 weeks after the first dose. The influenza vaccines will contain the three influenza virus strains chosen by the FDA. Each subject will receive by nasal spray a 0.2 ml dose (0.1 ml in each nostril) of the LAIV or 0.5 ml intramuscularly.

The duration of each study year is approximately five to ten months, from the time of enrollment (August to January, at the discretion of the investigators) depending on vaccine availability and the timing of influenza activity, to the end of the influenza season (May).

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent form by adult participant or parent/ legal guardian who are able to understand and comply with the protocol and assent when appropriate (usually age greater than or equal to 7 years)
* healthy subject, 4 through 18 years of age and none of the exclusion criteria

Exclusion Criteria:

* history of hypersensitivity, especially anaphylactic reaction, to any components of FluMist™, including eggs or egg products
* on aspirin therapy or aspirin-containing therapy
* history of Guillain-Barré syndrome
* known or suspected immune deficiency diseases such as combined immunodeficiency, agammaglobulinemia, and thymic abnormalities and conditions such as human immunodeficiency virus infection, malignancy, leukemia or lymphoma
* on immunosuppressive therapies such as systemic corticosteroids, alkylating drugs, antimetabolites, or radiation
* close contact within 21 days after vaccination with immunocompromised individuals
* history of asthma or reactive airway disease
* history of chronic or underlying diseases for which the licensed inactivated flu vaccine (IIV-T) is recommended such as chronic disorders of the cardiovascular and pulmonary systems, or chronic conditions such as metabolic diseases, renal dysfunction or hemoglobinopathies that required medical follow-up or hospitalization during the preceding year
* concurrent use with an anti-influenza compound
* pregnant or plans to become pregnant within 42 days after vaccination
* nursing mother and
* any condition which, in the opinion of the investigator, interferes with evaluation of the vaccine

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 29255 (Actual)
Dates: Start 1998-10 (Actual); Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro A Piedra, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Scott & White Hospital and Clinic, Temple, Texas
  - Scott & White Hospital and Clinic, Waco, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gaglani MJ, Piedra PA, Riggs M, Herschler G, Fewlass C, Glezen WP. Safety of the intranasal, trivalent, live attenuated influenza vaccine (LAIV) in children with intermittent wheezing in an open-label field trial. Pediatr Infect Dis J. 2008 May;27(5):444-52. doi: 10.1097/INF.0b013e3181660c2e. PMID 18401289
- [Result] Piedra PA, Gaglani MJ, Kozinetz CA, Herschler GB, Fewlass C, Harvey D, Zimmerman N, Glezen WP. Trivalent live attenuated intranasal influenza vaccine administered during the 2003-2004 influenza type A (H3N2) outbreak provided immediate, direct, and indirect protection in children. Pediatrics. 2007 Sep;120(3):e553-64. doi: 10.1542/peds.2006-2836. Epub 2007 Aug 13. PMID 17698577
- [Result] Halloran ME, Piedra PA, Longini IM Jr, Gaglani MJ, Schmotzer B, Fewlass C, Herschler GB, Glezen WP. Efficacy of trivalent, cold-adapted, influenza virus vaccine against influenza A (Fujian), a drift variant, during 2003-2004. Vaccine. 2007 May 16;25(20):4038-45. doi: 10.1016/j.vaccine.2007.02.060. Epub 2007 Mar 12. PMID 17395338
- [Result] Piedra PA, Gaglani MJ, Riggs M, Herschler G, Fewlass C, Watts M, Kozinetz C, Hessel C, Glezen WP. Live attenuated influenza vaccine, trivalent, is safe in healthy children 18 months to 4 years, 5 to 9 years, and 10 to 18 years of age in a community-based, nonrandomized, open-label trial. Pediatrics. 2005 Sep;116(3):e397-407. doi: 10.1542/peds.2004-2258. PMID 16140685
- [Result] Piedra PA, Gaglani MJ, Kozinetz CA, Herschler G, Riggs M, Griffith M, Fewlass C, Watts M, Hessel C, Cordova J, Glezen WP. Herd immunity in adults against influenza-related illnesses with use of the trivalent-live attenuated influenza vaccine (CAIV-T) in children. Vaccine. 2005 Feb 18;23(13):1540-8. doi: 10.1016/j.vaccine.2004.09.025. PMID 15694506
- [Result] Gaglani MJ, Piedra PA, Herschler GB, Griffith ME, Kozinetz CA, Riggs MW, Fewlass C, Halloran ME, Longini IM Jr, Glezen WP. Direct and total effectiveness of the intranasal, live-attenuated, trivalent cold-adapted influenza virus vaccine against the 2000-2001 influenza A(H1N1) and B epidemic in healthy children. Arch Pediatr Adolesc Med. 2004 Jan;158(1):65-73. doi: 10.1001/archpedi.158.1.65. PMID 14706961
- [Result] Halloran ME, Longini IM Jr, Gaglani MJ, Piedra PA, Chu H, Herschler GB, Glezen WP. Estimating efficacy of trivalent, cold-adapted, influenza virus vaccine (CAIV-T) against influenza A (H1N1) and B using surveillance cultures. Am J Epidemiol. 2003 Aug 15;158(4):305-11. doi: 10.1093/aje/kwg163. PMID 12915495
- [Derived] Glezen WP, Gaglani MJ, Kozinetz CA, Piedra PA. Direct and indirect effectiveness of influenza vaccination delivered to children at school preceding an epidemic caused by 3 new influenza virus variants. J Infect Dis. 2010 Dec 1;202(11):1626-33. doi: 10.1086/657089. Epub 2010 Oct 28. PMID 21028955

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants in the intervention cities were enrolled to the study and signed informed consent. The participants in the comparison cities were not enrolled to the study and the relevant data for these participants were obtained from the Scott and White Clinic database.
Groups:
- Intervention Cities: Eligible children 4 years of age and older whose parents provided consent (assent for children>7 years) in the intervention cites (Temple, Belton, Academy, Troy, Salado, Rogers, and Holland) were offered live attenuated or inactivated influenza vaccines through a school-based research vaccination program.
Period: Overall Study
Arm/Group | Intervention Cities
Started | 29255
Completed | 29255
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention Cities: Eligible children 4 years of age and older in the intervention cites (Temple, Belton, Academy, Troy, Salado, Rogers, and Holland with be offered live attenuated or inactivated influenza vaccines through a school-based research vaccination program.
Arm/Group | Intervention Cities
Number analyzed (Participants) | 29255
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 29255
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 8 [5 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15106
  Male | 14149
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9163
  Not Hispanic or Latino | 20092
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 203
  Asian | 519
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2335
  White | 24699
  More than one race | 1499
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 29255

OUTCOME MEASURES:

1. Primary Outcome: MAARI Rate During the Epidemic Period (2007-2008)
Description: The rate of MAARI (MAARIs/1000 persons-week) were compared between the intervention and comparison cities during the epidemic period (irrespective of the vaccination status). This data was obtained from the SWHP database.
Time Frame: 12/16/2007 to 3/29/2008 (15 weeks)
Population: Overall rate of MAARI (MAARIs/1000 persons-week) were compared between the intervention and comparison cities during the epidemic period (irrespective of the vaccination status). Total number of participants reflect the number of SWHP participants in the intervention and comparison cities respectively.
Measure: Number; unit: Number of MAARI
Units Other Than Participants: Person Weeks
Groups:
- Intervention Cities: Eligible children 4 years of age and older in the intervention cites (Temple, Belton, Academy, Troy, Salado, Rogers, and Holland were offered live attenuated or inactivated influenza vaccines through a school-based research vaccination program. Age-specific rates for medically attended acute respiratory illness (MAARI) in the influenza outbreak periods.
- Comparison Cities: Children living in the comparison cities (Waco, Bryan and College Station) which are within 90 miles of the intervention cites received their influenza vaccines by the local healthcare providers. Age-specific rates for medically attended acute respiratory illness (MAARI) in the influenza outbreak periods.
Arm/Group | Intervention Cities | Comparison Cities
Number analyzed (Participants) | 50665 | 67036
Number analyzed (Person Weeks) | 759975 | 1005540
Number of MAARI | 12503 | 18998
Statistical Analysis 1: Comparison: Intervention Cities vs Comparison Cities; Overall Effectiveness against MAARI during the Epidemic Period (2007-2008); Test type: Other; Incidence Rate Ratio = 0.89, 95% CI 2-sided [0.87 to 0.91]

2. Primary Outcome: MAARI Rate During the Epidemic Period (2008-2009)
Description: as for outcome 1
Time Frame: 1/4/2009 to 3/21/2009 (11 weeks)
Population: as for outcome 1
Measure: Number; unit: Number of MAARI
Units Other Than Participants: Person Weeks
Arm/Group | Intervention Cities | Comparison Cities
Number analyzed (Participants) | 50597 | 64969
Number analyzed (Person Weeks) | 556567 | 714659
Number of MAARI | 6630 | 12429
Statistical Analysis 1: Comparison: Intervention Cities vs Comparison Cities; Overall Effectiveness against MAARI during the Epidemic Period (2008-2009); Test type: Other; Incidence Rate Ratio = 0.69, 95% CI 2-sided [0.67 to 0.71]

3. Primary Outcome: MAARI Rate During the Epidemic and Pandemic Period (2009-2010)
Description: as for outcome 1
Time Frame: 8/25/09 to 4/3/10 (32 weeks)
Population: as for outcome 1
Measure: Number; unit: Number of MAARI
Units Other Than Participants: Person Weeks
Arm/Group | Intervention Cities | Comparison Cities
Number analyzed (Participants) | 44610 | 56052
Number analyzed (Person Weeks) | 1427521 | 1793665
Number of MAARI | 15155 | 25984
Statistical Analysis 1: Comparison: Intervention Cities vs Comparison Cities; Overall Effectiveness against MAARI during the Epidemic Period (2008-2009); Test type: Other; Incidence Rate Ratio = 0.75, 95% CI 2-sided [0.73 to 0.76]

4. Secondary Outcome: Proportion of SAEs Detected in LAIV Recipients
Description: Serious adverse events (SAEs) within 42 days post-LAIV vaccination will be captured in seasonal and pandemic vaccinated study subjects.
Time Frame: pre-, post- influenza vaccination
Population: This analyses was limited to the children enrolled in the intervention cities. 29255 doses of LAIV were administered to children 4-18 years of age. 21555 doses were seasonal LAIV and 7700 doses were pandemic LAIV.
Measure: Number; unit: proportion of events
Groups:
- Influenza Vaccine: Eligible children 4 years of age and older in the intervention cites (Temple, Belton, Academy, Troy, Salado, Rogers, and Holland) were offered live attenuated or inactivated influenza vaccines through a school-based research vaccination program. Serious adverse events (SAEs) and MAARI adverse events within 42 days post-LAIV vaccination were captured in seasonal and pandemic LAIV vaccinated study subjects in the intervention area.
Arm/Group | Influenza Vaccine
Number analyzed (Participants) | 29255
proportion of events
  Incidence of SAEs among seasonal LAIV recipients | 0.00005
  Incidence of SAEs among pandemic LAIV recipients | 0.00012

ADVERSE EVENTS:
Description: Non-serious adverse events were not captured during the course of this study except for pregnancy(ies).
Groups:
- All Enrolled Study Participants: Children 4 years of age and older in the intervention cites (Temple, Belton, Academy, Troy, Salado, Rogers, and Holland) with be offered live attenuated or inactivated influenza vaccines through a school-based research vaccination program. Children living in the comparison cities (Waco, Bryan and College Station) which are within 90 miles of the intervention cites will received their influenza vaccines (live attenuated or inactivated influenza vaccines) by the local healthcare providers
Arm/Group | All Enrolled Study Participants
Serious Adverse Events (participants affected / at risk) | 57/29255
Other Adverse Events (participants affected / at risk) | 1/29255
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Enrolled Study Participants (N=29255)
Psychiatric Disorder (Psychiatric disorders) | 3
Trauma/Skeletal Pain (Musculoskeletal and connective tissue disorders) | 2
Migraine/Headache (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 2
Elective Surgery (Investigations) | 5
Soft tissue and/or bone infection (Musculoskeletal and connective tissue disorders) | 2
Urinary Tract Infection (Renal and urinary disorders) | 1
Sepsis (General disorders) | 1
Meningitis (Nervous system disorders) | 2
Pharyngitis/Group A Strep/Abscess (Gastrointestinal disorders) | 1
Lower Respiratory Tract Infection (LRTI) (Respiratory, thoracic and mediastinal disorders) | 7
2009 H1N1 Pneumonia/LRTI (Respiratory, thoracic and mediastinal disorders) | 6
Acute Asthma Attack (Respiratory, thoracic and mediastinal disorders) | 2
Sickle Cell Crisis (Blood and lymphatic system disorders) | 1
Gastroenteritis/Mesentric Adenitis (Gastrointestinal disorders) | 1
Emesis and Weight Loss (Gastrointestinal disorders) | 1
Appendicitis (Gastrointestinal disorders) | 10
Acute abdominal pain (Gastrointestinal disorders) | 1
Intussususception (Gastrointestinal disorders) | 1
Henoch-Schonlein Purpura (Blood and lymphatic system disorders) | 1
Optic neuritis (Eye disorders) | 1
Guillain Barre Syndrom (Nervous system disorders) | 1
Oilgoarticular post-infectious arthritis (Musculoskeletal and connective tissue disorders) | 1
Death (General disorders) | 1
Carbon Monoxide Poisoning (General disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Enrolled Study Participants (N=29255)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No